CLINICAL TRIAL: NCT00465205
Title: A Randomized,Double-Blind , Placebo-Controlled Crossover Trial of Antivirals for Suppression of HSV and HIV Shedding in HIV-1, HSV-2 Co-infected Persons
Brief Title: HSV-2 Suppression to Reduce HIV-1 Levels in HIV-1 Co-infected Persons
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: GlaxoSmithKline (Industry); Asociación Civil Impacta Salud y Educación, Peru (Other)
Responsible Party: Connie Celum MD MPH, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 21760-A (2); AI277S7;AI38858;AI30731
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: HIV Infections; Herpes Simplex; Sexually Transmitted Diseases
Keywords: HIV infection; HIV Shedding; HSV suppression; Co-infected; Women; Reactivation; Valacyclovir; Treatment Naive
MeSH Terms: conditions — HIV Infections; Herpes Simplex; Sexually Transmitted Diseases | interventions — Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- I (Experimental)
  Interventions: Drug: Valacyclovir; Drug: Matching Placebo

INTERVENTIONS:
Drug: Valacyclovir — 500mg oral twice daily
  Other Names: Valtrex
Drug: Matching Placebo — 500 mg oral twice daily
  Other Names: Placebo for Valacyclovir

SUMMARY:
Over 80% of HIV-1 infected persons are also seropositive for HSV-2. Increasingly, clinical and epidemiologic evidence show the role of HSV in increasing HIV infectiousness. The evidence suggests that HSV is an important co-factor in HIV transmission.

The trial's purpose is to assess the reduction in HIV systemic and mucosal replication associated with valacyclovir for suppression of HSV-2 reactivation.

This randomized, double-blind, placebo controlled crossover trial of 20 HIV/HSV-2 co-infected women assessed the effects of daily valacyclovir on HIV-1 levels in blood and body fluids.

DETAILED DESCRIPTION:
Conducted in Lima Peru, 20 HIV-1 and HSV-2 seropositive women with CD4 counts greater than 200 and on no antiretroviral therapy were randomly assigned to receive valacyclovir 500 mg bid or placebo for the first 8 weeks of the study. After these 8 weeks, a 2-week washout period followed, which was then followed by the alternative regimen for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years old woman,
* Documented HIV-1 seropositive,
* CD4 count greater than 200,
* Not on HIV antiretroviral therapy,
* HSV-2 seropositive as determined by Focus EIA (IN >3.5)
* Not intending to move out of the area for the duration of study participation.
* Willing and able to:provide independent written informed consent;undergo clinical evaluations;take study drug as directed;adhere to follow-up schedule.
* Bacterial STDs (symptomatic STD syndromes or laboratory-confirmed asymptomatic gonorrhea and syphilis) are treated within two weeks of study enrollment and random assignment.

Exclusion Criteria:

Women who meet any of the following criteria are not eligible for this study:

* Known history of adverse reaction to valacyclovir, acyclovir or famciclovir;
* Planned open label use of acyclovir, valacyclovir, or famciclovir
* Known medical history of seizures
* Known renal failure, serum creatinine >2.0mg/dl
* Hematocrit < 30 %

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-01; Primary Completion 2005-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Plasma HIV-1 levels and HIV-1 mucosal shedding | 18 weeks

SECONDARY OUTCOMES:
Mucosal HSV-2 shedding | 18 weeks
Determine the temporal pattern of HIV shedding with respect to HSV-1 and HSV-2 reactivation; | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Connie Celum, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Asociacion Civil Impacta Salud y Educacion, Lima, Peru

REFERENCES:
- [Derived] Baeten JM, Strick LB, Lucchetti A, Whittington WL, Sanchez J, Coombs RW, Magaret A, Wald A, Corey L, Celum C. Herpes simplex virus (HSV)-suppressive therapy decreases plasma and genital HIV-1 levels in HSV-2/HIV-1 coinfected women: a randomized, placebo-controlled, cross-over trial. J Infect Dis. 2008 Dec 15;198(12):1804-8. doi: 10.1086/593214. PMID 18928378